CLINICAL TRIAL: NCT04196673
Title: Posterior Capsule Opafication of Two Different Hydrophobic Acrylic Intraocular Lenses: Vivinex iSert P261 vs. Acrysof SN60WF
Brief Title: Posterior Capsule Opafication of Two Different Hydrophobic Acrylic Intraocular Lenses
Acronym: Acryvivi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Clinical Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1560/2014
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Age Related Cataracts

STUDY DESIGN:
Intervention Model Description: The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. Cataract surgery with precedent bilateral randomized IOL implantation will be performed in subjects who have signed an informed consent form. Postoperative examinations will be implemented in accordance with the approved Investigational Plan on subjects and includes: visual acuity, slitlamp examination, fibrosis, posterior capsule opacification (PCO) score and YAG capsulotomy rate.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcon SN60WF (Experimental): Implantation of an intraocular lens Alcon SN60WF
  Interventions: Device: Alcon SN60WF
- Hoya Vivinex (Experimental): Implantation of an intraocular lens Hoya Vivinex
  Interventions: Device: Hoya Vivinex

INTERVENTIONS:
Device: Alcon SN60WF — Implantation of an intraocular lens Alcon SN60WF
  Arms: Alcon SN60WF
Device: Hoya Vivinex — Implantation of an intraocular lens Hoya Vivinex
  Arms: Hoya Vivinex

SUMMARY:
On the day of surgery, the first eye to be operated is randomised to receive a Vivinex , HOYA Surgical Optics GmbH or an SN60WF, Alcon, Fort Worth, Texas. The second eye to be operated receives the other IOL type.

A complete biomicroscopic examination, visual acuity testing using autorefractometer, contrast sensitivity testing, and standardised retroillumination photography for PCO evaluation, will be performed 6 month (30-60 days), 1.5 years (± 3 months) and 3 (± 3 months) years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract for which phacoemulsification extraction and posterior IOL implantation has planned
* Age 50 and older
* Visual potential in both eyes of 20/30 or better as determined by investigators estimation
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Preceding intraocular surgery or ocular trauma
* Relevant other ophthalmic diseases (such as pseudoexfoliation, glaucoma, uveitis, retinal degenerations, etc.)
* Laser treatment
* Uncontrolled systemic or ocular disease
* Infectious disease
* Pregnancy/Nursing

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-06-19 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
PCO score | 3 years
  subjectively and objectively graded: 0-10 (0= no PCO, 10= maximum PCO)

SECONDARY OUTCOMES:
Visual Acuity | 3 years
  UCDVA(uncorrected distance visual acuity), BCDVA (best corrected distance visual acuity)
Fibrosis | 3 years
  grade of fibrosis assessed subjectively at the slitlamp (grade 0=no fibrosis, grade 3=maximum fibrosis)
Subjective glistening score | 3 years
  neg, <10, 10-20, 20-30, 30-40, >40 uniform or localized
YAG capsulotomy rate | 3 years
  described subjectively at the slitlamp: was a YAG capsulotomy performed yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Menapace, Prof. Dr., Principal Investigator — Medical University of Vienna

IPD SHARING:
Plan to Share IPD: No